CLINICAL TRIAL: NCT00966628
Title: The Effect of Hypertonic Sodium Lactate on sVCAM-1 Level as a Surrogate Marker of Endothelial Capillary Leakage in Pediatric Dengue Shock Syndrome Patients
Brief Title: Effect of Hypertonic Sodium Lactate on sVCAM-1 Level as Surrogate Marker of Endothelial Capillary Leakage in Pediatric Dengue Shock Syndrome Patients (DSS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Innogene Kalbiotech Pte. Ltd (Industry)
Responsible Party: Dr. Rikrik Ilyas, Innogene Kalbiotech Pte. Ltd., Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006/IGK-KAL/08
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Dengue Shock Syndrome
Keywords: pediatric; dengue; hypertonic sodium lactate; fluid resuscitation; Ringer's lactate
MeSH Terms: conditions — Severe Dengue; Dengue | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ringer's lactate (Active Comparator)
  Interventions: Drug: Ringer's lactate
- Hypertonic sodium lactate (Experimental)
  Interventions: Drug: Hypertonic sodium lactate

INTERVENTIONS:
Drug: Hypertonic sodium lactate — Hypertonic sodium lactate 5 ml/kg BW administered within 15 minutes to restore hemodynamic status. If shock state did not recover with first infusion, study solution infused again at same dose. After recovery from shock state, patients receive maintenance dose at 1 mL/kgBW/hour for 12 hours. After 12 hr. infusion with study fluid, patients receive RL infusion as per standard protocol of DSS management at site.In case of repeated shock within 12 hours, study drugs can be infused again. If patient still not recovered from shock state, the patients will be given HES (Hydroxy-Ethyl Starch) infusion at dose of 20 mL/kgBW/15-30 min with maximum dose of 50 mL/kgBW/24 hours.
  Other Names: Totilac™
  Arms: Hypertonic sodium lactate
Drug: Ringer's lactate — Ringer lactate infused at dose 20 mL/kgBW within 15 minutes to restore hemodynamic status. If shock state did not recover with first infusion, study fluid infused again at same dose. After recovery from shock, patient received maintenance dose of RL. In case of repeated shock, patients received HES (Hydroxy-Ethyl Starch) infusion at dose of 20 mL/kgBW/15-30 min with maximum dose of 50 mL/kgBW/24 hours.
  Arms: Ringer's lactate

SUMMARY:
Dengue hemorrhagic fever (DHF) and dengue shock syndrome (DSS) are among the leading causes of pediatric hospitalization in Asia.Mortality rates range from 1% at centres experienced in fluid resuscitation, to upto 44% in established shock.The mainstay of DSS treatment is prompt, vigorous fluid resuscitation with isotonic crystalloid solutions, followed by plasma or colloid solutions for profound or continuing shock. However, this administration is often associated with fluid overload and induces edema in these patients.

Hence, we planned a parallel, randomized controlled trial comparing the efficacy and safety of solution containing half molar sodium lactate (Totilac™) with standard treatment(isotonic crystalloid Ringer's Lactate) in pediatric Dengue Shock Syndrome patients, using plasma soluble Vascular Cell Adhesion Molecule(sVCAM-1) levels as an indicator.

Hypertonic solutions restore hemodynamic status rapidly with increased cardiac performance and improved tissue perfusion. This is obtained with much smaller volumes.We plan to assess the efficacy and safety of hypertonic sodium lactate in resuscitation of DHF/DSS patients.

DETAILED DESCRIPTION:
Dengue affects an estimated 100 million people worldwide annually and is endemic in parts of Asia and the Americas, with increased incidence reported from many tropical countries recently.Dengue hemorrhagic fever (DHF) and dengue shock syndrome (DSS) are among the leading causes of pediatric hospitalization in Asia.Mortality rates range from 1% at centres experienced in fluid resuscitation, to upto 44% in established shock.

The mainstay of DSS treatment is prompt, vigorous fluid resuscitation with isotonic crystalloid solutions, followed by plasma or colloid solutions for profound or continuing shock. If appropriate volume resuscitation is started at an early stage, DSS is usually reversible. Patients who do not receive a proper treatment usually die within 12-24 hours after shock ensues. However, this administration is often associated with fluid overload and induces edema in these patients.

During hypovolemia in DHF/DSS, systemic hemodynamics and microcirculation are impaired, subsequently triggering a vicious cycle of progressive tissue damage that finally may lead to development of multiple organ failure. By adequately restoring intravascular volume, organ perfusion may be guaranteed, nutritive microcirculatory flow may be improved, and activation of a complex series of damaging cascades may be avoided.A solution that can rapidly restore systemic hemodynamic and improve microcirculation may be more beneficial in DHF/DSS patients.

Hypertonic solutions restore hemodynamic status rapidly with increased cardiac performance and improved tissue perfusion indicated by better urine output and tissue oxygenation. This is obtained with much smaller volumes.High lactate contained in hypertonic sodium lactate also functions as an alternate energy substrate.

However, the effects of hypertonic solution for resuscitating DHF/DSS patients have not yet investigated.Hence, we planned a parallel, randomized controlled trial comparing the efficacy and safety of solution containing half molar sodium lactate (Totilac™) with standard treatment(isotonic crystalloid Ringer's Lactate) in resuscitating pediatric Dengue Shock Syndrome patients, using plasma soluble Vascular Cell Adhesion Molecule(sVCAM-1) levels as an indicator of capillary endothelial leakage, which frequently occurs in DHF/DSS.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with dengue shock syndrome
* Ages 2-14 years
* Resuscitation treatment naïve for DSS
* Fulfill WHO criteria for dengue shock syndrome
* Signed informed consent

Exclusion Criteria:

* Patients with history of nephritic syndrome or severe renal impairment (creatinine > 2 mg/dL ), severe liver impairment (SGOT & SGPT > 2x normal), chronic diarrhea, severe malnutrition, diabetes mellitus, and history of hematological disorder based on anamnesis, physical examination, and/or lab exam.
* Patients who are confirmed to have suffered viral or bacterial infection based on anamnesis, physical examination, and lab exam

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of solution containing half molar sodium lactate (Totilac™) infusion on the plasma sVCAM-1 level | sVCAM-1 levels measured before resuscitation, after 6 hours, 12 hours, 24 hours & 48 hours post resuscitation

SECONDARY OUTCOMES:
To assess the effect of solution containing half molar sodium lactate (Totilac™) infusion on other efficacy and safety parameters | Hemodynamic parameters monitored hourly. Lab parameters measured 1 hour post resuscitation and every 3 hours thereafter, based on disease severity, upto 12 hours post resuscitation. Serology exams also done at day 5 from fever onset or thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Leverve, MD, PhD, Study Chair — INSERM-E0221-Bioenergetique Fondamentale et Appliquée Université Joseph Fourier, France; Dadang H Somasetia, SpA(K), MKes, Principal Investigator — Hasan Sadikin Hospital, Dept. of Pediatrics, Bandung, Indonesia
Locations (1):
- Hasan Sadikin Hospital, Dept. of Pediatrics, Bandung, West Java, Indonesia

REFERENCES:
- [Background] Ampaiwan Chuansumrit, MD & Kanchana Tangnararatchakit, MD, Pathophysiology and management of dengue hemorrhagic fever, Journal Compilation, 2006. Transfusion Alternatives in Transfusion Medicine 8 (Suppl. 1), 3-11
- [Background] Murgue B, Cassar O, Deparis X. Plasma concentrations of sVCAM-1 and severity of dengue infections. J Med Virol. 2001 Sep;65(1):97-104. PMID 11505450
- [Background] Wills BA, Nguyen MD, Ha TL, Dong TH, Tran TN, Le TT, Tran VD, Nguyen TH, Nguyen VC, Stepniewska K, White NJ, Farrar JJ. Comparison of three fluid solutions for resuscitation in dengue shock syndrome. N Engl J Med. 2005 Sep 1;353(9):877-89. doi: 10.1056/NEJMoa044057. PMID 16135832
- [Background] Bethell DB, Gamble J, Pham PL, Nguyen MD, Tran TH, Ha TH, Tran TN, Dong TH, Gartside IB, White NJ, Day NP. Noninvasive measurement of microvascular leakage in patients with dengue hemorrhagic fever. Clin Infect Dis. 2001 Jan 15;32(2):243-53. doi: 10.1086/318453. Epub 2001 Jan 15. PMID 11170914
- [Background] Schierhout G, Roberts I. Fluid resuscitation with colloid or crystalloid solutions in critically ill patients: a systematic review of randomised trials. BMJ. 1998 Mar 28;316(7136):961-4. doi: 10.1136/bmj.316.7136.961. PMID 9550953
- [Background] Gubler DJ. Dengue and dengue hemorrhagic fever. Clin Microbiol Rev. 1998 Jul;11(3):480-96. doi: 10.1128/CMR.11.3.480. PMID 9665979
- [Background] Jiang G, Klein JD, O'Neill WC. Growth factors stimulate the Na-K-2Cl cotransporter NKCC1 through a novel Cl(-)-dependent mechanism. Am J Physiol Cell Physiol. 2001 Dec;281(6):C1948-53. doi: 10.1152/ajpcell.2001.281.6.C1948. PMID 11698253
- [Background] Boldt J. New light on intravascular volume replacement regimens: what did we learn from the past three years? Anesth Analg. 2003 Dec;97(6):1595-1604. doi: 10.1213/01.ANE.0000089961.15975.78. PMID 14633526 (Retraction: PMID 33031689 Anesth Analg. 2020 Aug;131(2):e137)
- [Background] Leverve XM, Boon C, Hakim T, Anwar M, Siregar E, Mustafa I. Half-molar sodium-lactate solution has a beneficial effect in patients after coronary artery bypass grafting. Intensive Care Med. 2008 Oct;34(10):1796-803. doi: 10.1007/s00134-008-1165-x. Epub 2008 Jun 18. PMID 18563389
- [Background] Leverve XM, Mustafa I. Lactate: A key metabolite in the intercellular metabolic interplay. Crit Care. 2002 Aug;6(4):284-5. doi: 10.1186/cc1509. Epub 2002 Jul 8. PMID 12225597
- [Background] Mustafa I, Leverve XM. Metabolic and hemodynamic effects of hypertonic solutions: sodium-lactate versus sodium chloride infusion in postoperative patients. Shock. 2002 Oct;18(4):306-10. doi: 10.1097/00024382-200210000-00003. PMID 12392272
- [Background] Valero N, Espina LM, Anez G, Torres E, Mosquera JA. Short report: increased level of serum nitric oxide in patients with dengue. Am J Trop Med Hyg. 2002 Jun;66(6):762-4. doi: 10.4269/ajtmh.2002.66.762. PMID 12224588
- [Background] Ngo NT, Cao XT, Kneen R, Wills B, Nguyen VM, Nguyen TQ, Chu VT, Nguyen TT, Simpson JA, Solomon T, White NJ, Farrar J. Acute management of dengue shock syndrome: a randomized double-blind comparison of 4 intravenous fluid regimens in the first hour. Clin Infect Dis. 2001 Jan 15;32(2):204-13. doi: 10.1086/318479. Epub 2001 Jan 15. PMID 11170909
- [Background] O'Neill WC. Physiological significance of volume-regulatory transporters. Am J Physiol. 1999 May;276(5):C995-C1011. doi: 10.1152/ajpcell.1999.276.5.C995. PMID 10329946
- [Background] Avirutnan P, Malasit P, Seliger B, Bhakdi S, Husmann M. Dengue virus infection of human endothelial cells leads to chemokine production, complement activation, and apoptosis. J Immunol. 1998 Dec 1;161(11):6338-46. PMID 9834124
- [Background] Rocha-e-Silva M, Poli de Figueiredo LF. Small volume hypertonic resuscitation of circulatory shock. Clinics (Sao Paulo). 2005 Apr;60(2):159-72. doi: 10.1590/s1807-59322005000200013. Epub 2005 Apr 26. PMID 15880253
- [Background] Lawn SD, Tilley R, Lloyd G, Finlayson C, Tolley H, Newman P, Rice P, Harrison TS. Dengue hemorrhagic fever with fulminant hepatic failure in an immigrant returning to Bangladesh. Clin Infect Dis. 2003 Jul 1;37(1):e1-4. doi: 10.1086/375601. Epub 2003 Jun 25. PMID 12830429
- [Background] Svensen CH. Hypertonic Solutions: An Update. ITACCS Clinical Issues. 2002, 6 -12
- [Background] Tan TS, Tan KH, Ng HP, Loh MW. The effects of hypertonic saline solution (7.5%) on coagulation and fibrinolysis: an in vitro assessment using thromboelastography. Anaesthesia. 2002 Jul;57(7):644-8. doi: 10.1046/j.1365-2044.2002.02603.x. PMID 12059821
- [Background] World Health Organization, Dengue, Dengue Haemorrhagic Fever and Dengue Shock Syndrome in the Context of the Integrated Management of Childhood Illness, 2005
- [Derived] Somasetia DH, Setiati TE, Sjahrodji AM, Idjradinata PS, Setiabudi D, Roth H, Ichai C, Fontaine E, Leverve XM. Early resuscitation of dengue shock syndrome in children with hyperosmolar sodium-lactate: a randomized single-blind clinical trial of efficacy and safety. Crit Care. 2014 Sep 5;18(5):466. doi: 10.1186/s13054-014-0466-4. PMID 25189175